CLINICAL TRIAL: NCT06006806
Title: Evaluation of Radiobiological Effects in Skin Toxicities for Breast Cancer Patients With Pencil Beam Scanning Proton Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Covenant Health Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-474 INV
Record Dates: First submitted 2023-08-14; First posted 2023-08-23 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Stage I
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The goal of this study is to measure skin reactions during proton therapy for 100 patients over a period of three years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Radiation: Pencil Beam Scanning Proton Therapy — Part of the normal proton therapy process is to have a CT scan (called a CT simulation) performed that is used to create a proton treatment plan. A proton treatment plan is a computer model of the proton beam that is used to calculate where the protons will go inside the body. During the treatment planning process, the clinical team works to find the best possible placement of the protons. This study uses a process called "Spot Delete" to keep protons from stopping in the skin, which is believed to be related to skin reddening. Spot Delete is a software application that was developed at the Thompson Proton Center and is used in the treatment planning process.
  Other Names: Spot Delete

SUMMARY:
This purpose of this study is to examine skin reactions (called radiation dermatitis) that occur during pencil beam scanning (PBS) proton therapy. The researchers will test a unique technique called "Spot Delete" to see if it can reduce skin reactions for breast patients treated with PBS. They will also use a special computer model to study how the energy of the proton beam (linear energy transfer) is related to these skin reactions. The study involves creating a treatment plan based on a CT scan, which helps guide the proton beam in the body. The clinical team uses this CT scan to find the best placement for the protons. The "Spot Delete" method prevents protons from stopping in the skin, which is thought to cause skin redness.

DETAILED DESCRIPTION:
During the study, digital photos of patients' skin will be taken to assess the amount of redness, without revealing their identity. Patients will be given a self-report questionnaire and medical staff will document the skin reactions in the patients' medical charts. The degree of skin reactions will be compared against historical occurrence rates, and the location of any skin reactions that occur will be compared against the predicted location from the computer model. In this study, we aim to test the hypothesis that the "Spot Delete" technique in proton therapy reduces radiation dermatitis in breast cancer patients compared to historical data from patients who underwent regular proton therapy without the technique. To evaluate this, we will compare the extent of skin reactions in patients who receive proton therapy with the "Spot Delete" technique to historical data from patients who did not receive this treatment.

The effectiveness of the technique will be evaluated by measuring and documenting the degree of skin reactions in patients undergoing proton therapy with the Spot Delete technique. Digital photographs of the treatment area will be taken to assess radiation dermatitis using the treatment using the Common Terminology Criteria for Adverse Events (CTCAE) ver. 5.0 and using the Radiation Dermatitis Severity (RDS) scoring system. Radiation dermatitis will be assessed at baseline, weekly after every fifth treatment session, at the end of treatment, and at 2 post treatment follow-up appointments (e.g. 1-month and 6-months post treatment).These results will be compared to historical occurrence rates of skin reactions in regular proton therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have signed an approved consent form conforming to federal and institutional guidelines.
* Patients must be equal to or greater than 18 years old.
* The patient must have stage 0, I, II, or III breast cancer
* On histological examination, the tumor must be ductal carcinoma in-situ (DCIS) or invasive adenocarcinoma of the breast
* Surgical treatment of the breast must have been lumpectomy or mastectomy
* Patients must have an estrogen receptor (ER) analysis performed on the primary tumor
* Progesterone (PgR) analysis is desired but not mandatory
* No serious health conditions as determined by physician that would impact ability to complete treatment or impact skin in the area of treatment

Exclusion Criteria:

* Stage IV breast cancer
* Non-epithelial breast malignancies such as sarcoma or lymphoma
* Paget's disease of the nipple
* Prior breast or thoracic radiation therapy (RT) for any condition.
* Collagen vascular disease, specifically dermatomyositis with a Creatine phosphokinase (CPK) level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
* Pregnancy or lactation
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men are not eligible for this study
Enrollment: 100 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2028-07-07 (Estimated); Study Completion 2030-07-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in Radiation Dermatitis | weekly assessments over 10 weeks
  "Spot Delete" technique in proton therapy reduces radiation dermatitis in breast cancer patients compared to historical data from patients who underwent regular proton therapy without the technique. Assessed by photographs, questionnaires and assessment using CTCAE and Radiation Dermatitis Severity scoring system.

SECONDARY OUTCOMES:
linear energy transfer (LET) of the proton beam | LET calculated at treatment completion for each subject and then compared over the 10 weeks of assessment if radiation dermatitis or other skin reaction is reported. At that time data will be compared.
  A secondary objective of this study is to investigate how the linear energy transfer (LET) of the proton beam is related to skin reactions. , LET will be calculated using RayStation for each patient enrolled in the study. The skin reactions' location and severity will be compared with the calculated LET values, allowing researchers to determine any correlation between LET and skin reactions. In addition, the actual location of any skin reactions that occur during the study will be compared to the predicted location from the computer model

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Hedrick, PhD, Principal Investigator — Director of Medical Physics
Locations (1):
- Thompson Proton Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No